CLINICAL TRIAL: NCT07132710
Title: Strategy for Optimizing the Use of Virtual Reality by Reorganizing Practices
Brief Title: Reorganization Strategy to Optimize the Use of Virtual Reality
Acronym: S'OUVRIR
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_1241
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Adult Patients Managed in a Cardiac Critical Care Unit With a Pathology Requiring at Least One Potentially Painful and Anxiety-provoking Invasive Procedure
Keywords: Patient experience; virtual reality; critical care; job satisfaction; organizational innovation; qualitative study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- VR mask potential users in critical care: Patients and caregivers of cardiac critical care units likely to use a VR mask for therapeutic purposes
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — Patients and caregivers will be interviewed about the barriers and facilitators to the use of VR masks in the management of pain and anxiety, in order to propose organizational changes that encourage their use.

SUMMARY:
The benefits of virtual reality (VR) in managing pain and anxiety for critical care patients has never been demonstrated, even if a positive effect has been demonstrated in other populations of patients. A preliminary survey in 8 critical care units equipped with the VR mask, identified a under-use of masks by critical care teams. Before addressing the question of the effectiveness of the VR mask in a population of critical care patients, we must first identify the barriers and facilitators to its use and propose a new organization in critical care units promoting the use of VR mask by autonomous caregivers. A qualitative study will be conducted with patients and caregivers of a critical care unit to identify the barriers and facilitators to the use of virtual reality masks in the management of pain and anxiety by caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer caregivers working in the cardiac critical care unit for at least 6 months.
* Adult patients treated in the unit with a condition requiring at least one potentially painful and anxiety-provoking invasive procedure (e.g., Central Venous Line placement, Arterial Catheter Insertion, ...) allowing the use of the VR mask.
* Patients able to understand the instructions without language barriers, to ensure the validity of the interviews and the quality of the data collected.

Exclusion Criteria:

* Staff not volunteering to participate in the study.
* Patients whose condition presents a medical contraindication to the use of VR mask or who present cognitive disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As for the caregivers, the team is currently made up of 42 nurses and 35 care assitants, so our sample will be 12 nurses and 8 care assistants to be representative of the team.
  As for the patients,10 volunteer from the cardiac critical care unit who meet the eligibility criteria will be selected to ensure the greatest possible diversity of patient profiles.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Identify the barriers and facilitators to the use of virtual reality mask by paramedical staff in the management of invasive care for critical care patients | Participants will be interviewed once (about one-hour interview)
  Patients and caregivers of a cardiac critical care unit will be interviewed (semi-structured interviews) to gather their perceptions on the use of virtual reality mask for pain and anxiety management in invasive care for critical care patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel - Hospices Civils de Lyon, Bron, France, France